CLINICAL TRIAL: NCT03424226
Title: Sickness Evaluation at Altitude With Acetazolamide at Relative Dosages
Acronym: SEAWARD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Grant S Lipman, Associate Professor Department of Emergency Medicine, Stanford University, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 44765
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Acute Mountain Sickness
MeSH Terms: conditions — Altitude Sickness | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Visually identical pills
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- day of acetazolamide (Experimental): acetazolamide 125mg twice a day, started morning of ascent
  Interventions: Drug: Acetazolamide
- night before acetazolamide (Active Comparator): acetazolamide 125mg twice a day, started evening before ascent
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Acetazolamide — a diuretic and commonly used medication for prevention and treatment of acute mountain sickness
  Other Names: diamox

SUMMARY:
This double blind randomized trial will compare acetazolamide taken the morning of ascent to acetazolamide taken the evening prior to ascent for the prevention of acute mountain sickness (AMS). The day of ascent dosing has not been studied as a powered primary outcome. The study population is hikers who are ascending at their own rate under their own power in a true hiking environment at the White Mountain Research Station, Owen Valley Lab (OVL) and Bancroft Station (BAR), Bancroft Peak, White Mountain, California

DETAILED DESCRIPTION:
The specific aim of this study is to determine whether acetazolamide started the day-of ascent is inferior to the standard night before ascent dose of acetazolamide for the prevention of acute mountain sickness (AMS) in travelers in travelers to high altitude. Acetazolamide has been examined in over 200 high altitude studies over the past 50 years, and is the most commonly used drug for AMS prevention in the high mountains of Nepal, Western Europe, and Africa. Current Wilderness Medical Society Practice Guidelines recommend a 125mg dose of acetazolamide daily started the day or evening prior to ascent. However, day of ascent dosage has recently been found to be effective prophylaxis for severe AMS compared to placebo, but efficacy of day-of ascent dosage has not be confirmed versus standard acetazolamide dosage.

While acetazolamide is commonly used as an acclimatization aid, it is traditionally started the day or evening prior to ascent to theoretically optimize diuretic effect and compensatory respiratory changes. This timing may be impractical when rapid ascent is necessary, such as in search and rescue and military operations, or for the general recreationalists, trekkers, or climbers who do not have time to start prophylaxis prior to heading into the mountains. As there are an estimated 100 million recreationalists annually who ascend to high altitude around the world, innovation on optimal timing has a potentially large impact on traveler safety.

Acetazolamide has a time of onset between 60 - 90 minutes when taken as an immediate release tablet, with peak effect between 2 - 4 hours. With these pharmacokinetics in mind, we recently found that there was an observed robust protective effect of acetazolamide on severe AMS when taken the morning of ascent, and this was the first study to examine day-of dosing. This novel finding has not been otherwise investigated, and confirmation of this unique observation has the potential to increase acetazolamide'sits usage in "high risk" populations maximizing safety, while minimizing discomfort and poor sleep from pre-ascent nocturia., such as trekkers, skiers, climbers, and tactical missions requiring rapid ascents in the mountains of North America and Europe.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 healthy non-pregnant volunteer
* live at low elevation < 4000 ft
* Arrange your own transportation to WMRS (Bishop) by Friday evening of study weekend
* Available for full study duration (Friday PM-Sunday AM)

Exclusion Criteria:

* Age <18 or >75, Pregnant, Live at altitude >4000 ft Slept at altitude > 4000ft within 1 week of study Allergic to acetazolamide, sulfa drugs, Taking non-steroidal anti-inflammatory drugs, Acetazolamide, or Corticosteroids 1 week prior to study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-08-04 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
incidence of acute mountain sickness | 2 days
  incidence of acute mountain sickness by Lake Louise Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No